CLINICAL TRIAL: NCT00050375
Title: A Double-Blind, Placebo-Controlled, Multicenter Clinical Trial of Intravenous OvaRex® MAb-B43.13 as Post Chemotherapy Consolidation for Epithelial Carcinoma of Ovarian, Tubal or Peritoneal Origin
Brief Title: Clinical Trial for Ovarian Cancer (OvaRex®)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed by sponser
Sponsor: Unither Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OVA-Gy-17; NCT00068354 (obsolete NCT alias)
Record Dates: First submitted 2002-12-05; First posted 2002-12-06 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2006-06

CONDITIONS: Ovarian Cancer
Keywords: OvaRex; ovarian; CA125; murine; antibody; immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — oregovomab

INTERVENTIONS:
Drug: oregovomab

SUMMARY:
This study will compare the time to disease relapse between OvaRex® MAb-B43.13-treated patients and placebo-treated patients. This study will also compare assessments of survival, quality of life, immune response and safety between active and placebo groups.

DETAILED DESCRIPTION:
This a Phase III, double-blind, placebo-controlled, multi-center study of intravenous OvaRex® MAb-B43.13 as post-chemotherapy consolidation for epithelial carcinoma of ovarian, tubal, or peritoneal origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological diagnosis of epithelial adenocarcinoma of ovarian, tubal or peritoneal origin, and their disease is classified as FIGO Stage III or IV. Histological diagnosis must have been confirmed by site pathology review of slides as documented by the site investigator. These slides must be made available for sponsor review.
* Patients must have had an elevated serum CA125 level (per reference lab normal range) measured prior to or at surgery (i.e., not later than the immediate post-surgery period when the patient is in the surgical recovery room). If a pre-surgical CA125 measurement is not available, then the patient must have had: (a) a serum CA125 level ≥100 U/mL, and (b) tumor tissue that has been demonstrated by immunohistochemical methods to express CA125.
* Patients must have had a documented serum CA125 level ≤65 U/mL prior to the third cycle of front-line chemotherapy.
* Patients must have had microscopic or small diameter residual disease following primary de-bulking surgical procedure.
* Patients must have received chemotherapy that included a platinum compound and a taxane following appropriate staging procedures. Front-line treatment can include no more than 8 cycles of chemotherapy.
* Patients must have had a complete clinical response to their front-line surgery and chemotherapy. A complete clinical response is defined as one in which the patient had a normal physical examination, no conclusive evidence of residual tumor by CT of the abdomen and pelvis, a normal chest x-ray, and a serum CA125 level at least 5 U/mL but less than 35 U/mL as measured in the pretreatment baseline laboratories by the protocol Central Lab.
* Patients must have undergone no more than one interval de-bulking procedure.
* Patients must receive their first dose of study medication between 4 and 12 weeks after completing their last dose of front-line chemotherapy.
* Patients must have voluntarily agreed to participate and have signed the informed consent, and are willing to complete all study procedures.

Exclusion Criteria:

* Patients who have received more than one prior regimen of chemotherapy. A change in chemotherapy agents is permitted during the patient's primary therapy provided that the change is considered to be part of the initial chemotherapy treatment regimen.
* Patients with known refractory or recurrent epithelial adenocarcinoma of ovarian, tubal, or peritoneal origin requiring chemotherapy.
* Patients who have compromised hematopoietic function (hemoglobin <8.0 g/dL; lymphocyte count <300 mm³; neutrophil count <1000 mm³; platelet count <100,000 mm³.
* Patients with hepatic dysfunction defined as a bilirubin >1.5 times the upper normal limits, LDH, SGOT and SGPT>2 times upper limits of normal or albumin <3.5 g/dL.
* Patients with severe renal dysfunction defined as a serum creatinine >1.6 mg/dL.
* Patients with a known allergy to murine proteins or have had a documented anaphylactic reaction to any drug, or a known hypersensitivity to diphenhydramine or other antihistamines of similar chemical structure.
* Patients who have contraindications to the use of pressor agents.
* Patients being chronically treated with immunosuppressive drugs such as cyclosporin, ACTH, or systemic corticosteroids.
* Patients who have received immunotherapy (interferons, tumor necrosis factor, other cytokines [e.g., interleukins] or biological response modifiers, or BCG vaccines) within 6 weeks of receiving their first dose of study medication. Patients who have received hemopoietic factors are acceptable.
* Patients who have had a splenectomy.
* Patients with uncontrolled diseases other than cancer will be excluded. Patients with chronic diseases that are well controlled (e.g., diabetes mellitus, hypertension) are eligible.
* Patients who have a concurrent illness or chronically taking medication, which would confound the results of the study, preclude the patient from completing the study, or mask an adverse reaction.
* Patients who have a concurrent malignancy (except non-melanoma of the skin, in situ carcinoma of cervix), unless the patient received curative treatment and has been disease free for greater than or equal to 5 years.
* Patients receiving other investigational drugs within 30 days of enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354
Dates: Start 2002-12; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - Western Regional Community Clinical Oncology Program, Phoenix, Arizona
  - Little Rock Hematology Oncology Assoc., Little Rock, Arkansas
  - St. Jude Medical Center, Fullerton, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Gynecologic Oncology Associates, Newport Beach, California
  - University of California, Irvine, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford University, Stanford, California
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - University of Connecticut Cancer Center, Farmington, Connecticut
  - Northwestern Connecticut Oncology Hematology Associates, LLP, Torrington, Connecticut
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - H. Lee Moffitt Cancer Center and Research, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - The University of Chicago Hospitals, Chicago, Illinois
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Michiana Hematology Oncology PC, South Bend, Indiana
  - Brown Cancer Center, Louisville, Kentucky
  - Louisville Oncology, Louisville, Kentucky
  - Lake Charles Medical Surgical Clinic, Lake Charles, Louisiana
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - The Harry and Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - New England Medical Center, Boston, Massachusetts
  - Women's Specialty Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - SUNY-HSC Syracuse, Crouse Hospital, Syracuse, New York
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital - Health Systems, Cleveland, Ohio
  - GYN Oncology and Pelvic Surgery Associates, Columbus, Ohio
  - ProMedica Health Systems, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists-Northrup, Portland, Oregon
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University School of Medicine, Providence, Rhode Island
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Gynecologic Oncology Research and Development, Greenville, South Carolina
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - West Clinic, PC, Memphis, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Southwest Regional Cancer Center, Austin, Texas
  - Univ. of Texas SW Medical Center at Dallas, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VA Oncology Associates, Norfolk, Virginia
  - Carilion GYN Oncology Associates, Roanoke, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington